CLINICAL TRIAL: NCT03454360
Title: Collection of Specific Health And Patient Related Criteria Used to Select traNsapical TAVI Treatment and correspondinG outcomEs: CHANGE Neo™ TA Registry
Brief Title: CHANGE Neo™ TA Registry With ACURATE Neo™ Aortic Bioprosthesis and ACURATE Neo™ TA Transapical Delivery System
Status: Terminated | Type: Observational
Why Stopped: Sponsor business decision unrelated to product safety or efficacy.
Sponsor: Symetis SA (Industry)
Responsible Party: Sponsor
Organization: Boston Scientific Corporation (Industry)
Other Study IDs: 2016-03
Record Dates: First submitted 2017-07-31; First posted 2018-03-05 (Actual); Last update posted 2020-12-11 (Actual); Status verified 2020-12

CONDITIONS: Aortic Stenosis
Keywords: TAVI; Transcatheter Aortic Valve Replacement; Transcatheter Aortic Valve; Transapical Access
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: ACURATE neo™ Aortic Bioprosthesis — TAVI; Transcatheter Aortic Valve Replacement. Transapical Access.
  Other Names: ACURATE neo™ TA Delivery System

SUMMARY:
The purpose of this registry is to collect specific health and patient data to identify more precisely the patient population undergoing TA aortic valve replacement with the ACURATE neo™ Aortic biprosthesis and ACURATE neo™ TA Transapical Delivery System.

Safety and efficacy data will be collected to support the commercial use of the ACURATE neo™ Aortic Bioprosthesis and ACURATE neo™ TA Transapical Delivery System in a specific TA population.

As per IFU, the ACURATE neo™ and its ACURATE neo™ TA Delivery System are intended for use in minimally invasive, transcatheter aortic valve replacement using transapical access in patients presenting with severe aortic valve stenosis.

DETAILED DESCRIPTION:
The Primary Objective of this post-market registry is to collect specific health and patient characteristics to understand the indication for TA-TAVI and to further evaluate the safety and performance of the ACURATE neo ™ Aortic Bioprosthesis and ACURATE neo™ TA Transapical Delivery System in a specific TA population, consisting of 200 consented patients.

ELIGIBILITY:
Inclusion criteria:

* Symptomatic patients with severe aortic stenosis;
* Institution heart team determines that aortic valve replacement ACURATE neoTM device using its transapical delivery system is appropriate;

Exclusion criteria:

- Patients unable or unwilling to give inform consent;

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All subjects with severe aortic stenosis, for whom the transapical access is the most suitable approach as per heart-team consensus, who signed the Informed Consent Form (ICF) approved by the Independent Ethics Committee (IEC), and are deemed to be candidates to undergo transcatheter aortic valve implantation with the ACURATE neo™ Aortic Bioprosthesis and its Transapical Delivery System as per clinical practice at each participating site
Sampling Method: Non-Probability Sample
Enrollment: 107 (Actual)
Dates: Start 2018-02-06 (Actual); Primary Completion 2020-04-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
All cause mortality | 30 days
  the rate of all-cause mortality as measured at 30-days

SECONDARY OUTCOMES:
Safety and performance data will be collected to support the commercial use of the ACURATE neo ™ Aortic Bioprosthesis and ACURATE neo™ TA Transapical Delivery System in a specific TA population. | Procedure to Discharge, 30 days and 12-months
  Clinical events as defined per VARC 2 consensus document at procedure:
  All cause mortality; Stroke; Myocardial Infarction; Bleeding complication; Acute kidney injury; Vascular complication; Conduction disturbances and arrhythmia; Other TAVI-related complications
Procedural Success | Procedure to 24-hours
  Defined as absence of intra-procedure mortality (procedure to 24H) AND absence of complications arising during implantation of the prosthetic valve such as: inability to properly seat the valve in the annulus; need for more than one implanted aortic bioprosthesis (valve-in-valve or ectopic deployment) or if a surgical aortic valve replacement is required to correct a severe aortic regurgitation or procedure complication. The procedure can be considered as success despite the presence of residual aortic regurgitation, which may be due to the anatomic configuration of the annulus or a calcific valvular annulus.
Device Success | Post-procedure to Discharge.
  Defined as;
  * Absence of intra-procedure mortality (procedure to 24H) AND,
  * Correct positioning (placement in the annulus with no impairment of aortic bioprosthesis function) of a single prosthetic heart valve into the proper anatomical location AND,
  * Intended performance of the prosthetic heart valve assessed prior to discharge per local standard of care and defined as:
    * No prosthesis-patient mismatch (EAOi >0.85 cm2/m2 or EAOi >0.7 cm2/m2 for BMI ≥30 kg/m2) ) AND,
    * Mean aortic valve gradient <20mmHg or peak velocity < 3 m/s AND,
    * No moderate or severe prosthetic valve regurgitation.
  For echo parameters for the performance assessment, a pre-discharge echo examination should be performed as per local standard of care. If echo parameter pre-discharge is missing, any echo parameter within 45 days post-procedure may be used.
VARC 2 Composite Safety | 30-days
  Defined as:
  * All-cause mortality
  * All stroke
  * Life-threatening bleeding
  * Acute Kidney Injury- Stage 2 or 3
  * Coronary Artery Obstruction requiring intervention
  * Major Vascular Complications
  * Valve-related dysfunction requiring repeat procedure
Functional improvement as per NYHA Functional Classification | from baseline to, discharge, 30-days and 12-months follow-up.
  Change on NYHA Class between baseline and different follow-up
Improvement of EOA and mean Trans-prosthetic gradient | from baseline to discharge, 30- days and 12 months follow-up
  If the echo parameter pre-discharge is missing to assess the intended performance, any echo parameter data within 45-days post procedure may be used for the missing values;
Total Aortic Regurgitation | post-procedure, prior to discharge, at 30-days and 12-months follow-up;
  Change on Aortic Regurgitation over time at follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Michael Hilker, Prof.Dr.med, Principal Investigator — Universitätsklinikum Regensburg
Locations (10):
- Germany (10):
  - Kerckhoff Klinik, Bad Nauheim
  - Herz-und Gefäß-Kilink GmbH, Bad Neustadt an der Saale
  - Krankenhausbetriebgesellschaft, Bad Oeynhausen
  - BG Klinik Bergmannsheil, Bochum
  - Universitätsklinikum Frankfurt- Klinik für Thorax, Herz und thorakale Gefæßchirurgie, Frankfurt
  - Universitäts-Herzzentrum Freiburg-Bad Krozingen, Freiburg im Breisgau
  - Universitätsklinikum Hamburg-Eppendorf, Hamburg
  - Herzzentrum Leipzig, Leipzig
  - Deutsches Herzzentrum München, München
  - Universitätsklinikum Regensburg, Regensburg

IPD SHARING:
Plan to Share IPD: Undecided
The data and study protocol for this clinical trial may be made available to other researchers in accordance with the Boston Scientific Data Sharing Policy (http://www.bostonscientific.com/en-US/data-sharing-requests.html).